CLINICAL TRIAL: NCT04380623
Title: A Tailored, Health Communication Intervention for HPV Vaccine Hesitant Families
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meharry Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-12-890
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Human Papilloma Virus; HPV-Related Carcinoma; Vaccine Refusal; Parents; Program, Communication
MeSH Terms: conditions — Vaccination Refusal; Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Phone-Based Web-Page: HPV vaccine (Experimental): Parents who have already declined the HPV vaccine for their adolescent will receive pre-visit, tailored education information on the HPV vaccine via a text message with a website link.
  Interventions: Behavioral: Mobile Phone-Based Web-Page: HPV vaccine
- Mobile Phone-Based Web-Page: Healthy Lifestyles (Active Comparator): Parents who have already declined the HPV vaccine for their adolescent will receive pre-visit education information on an unrelated topic (e.g., healthy eating and physical activity) via a text message with a website link.
  Interventions: Behavioral: Mobile Phone-Based Web-Page: HPV vaccine

INTERVENTIONS:
Behavioral: Mobile Phone-Based Web-Page: HPV vaccine — Website to be accessed via mobile phone to deliver tailored educational material

SUMMARY:
The human papillomavirus (HPV) causes 90% of cervical cancers and is implicated in multiple other cancers. The HPV vaccine can prevent the vast majority of these cancers, but it is underused in adolescents, especially among those within vaccine hesitant (VH) parents. The proposed research is to develop and pilot test a tailored, health communication intervention aimed to increase HPV vaccination among VH parents. The proposed research is innovative because no evidence-based health communication interventions target HPV VH parents, and we will use stakeholder engagement throughout this study. The research will add knowledge on how tailored education provided before a doctor's visit can play a role in improving HPV vaccination rates among underserved, VH parents.

DETAILED DESCRIPTION:
The goal of this K01 application is to develop and pilot test an individually tailored, pre-visit health communication intervention targeting HPV-VH parents. The partnering clinic is Meharry Medical College Pediatric Group (MMC Pediatrics), a safety-net clinic serving primarily publicly-insured and uninsured patients. The study has three specific aims.

Aim 1. To develop a tailored, health communication intervention targeting HPV-VH parents prior to clinic visits. The tailored intervention will be delivered to VH parents via mobile phones. Investigators will draft initial content based on the Theory of Reasoned Action and Health Belief Model, previous VH research,14 and preliminary data. Then semi-structured interviews will be conducted with 25-30 VH parents who previously declined the HPV vaccine and 10 physicians to elicit feedback on draft content. Qualitative data will be collected and analyzed iteratively, informing successive modifications to the intervention to cover a range of potential concerns for VH parents, enhance message relevance, and refine the intervention delivery process. Next, investigators will work with MMC Pediatrics to develop and refine the study protocol. Investigators will pre-test and get feedback on the protocol from 16 VH parents and 3 physicians to maximize acceptance and feasibility.

Aim 2. Conduct a pilot study of the intervention and study protocol to demonstrate feasibility for the future full-scale randomized control trial (RCT). Based on Aim 1, investigators will conduct a small, pilot RCT with 70 VH parents with scheduled clinic visits. Feasibility indicators are recruitment rates, retention rates, and ability to ascertain patients' post-visit HPV vaccine status in the clinical record. VHealth software will be used to extract information from the EHR to identify potentially eligible patients with a previous HPV vaccine refusal and to determine the whether an HPV vaccine dose was received during the scheduled visit.

Aim 3. Examine acceptability of the intervention and protocol among parents and providers. Parents participating in the pilot study will complete a post-visit survey to measure acceptability of the intervention and protocol, provider trust/rapport, and satisfaction with provider-patient communication. In addition, investigators will conduct semi-structured debriefing interviews with a subset of 20-30 parents and 3 providers to gather qualitative data about their experiences (e.g., unforeseen problems and barriers) and their perceptions of acceptability of the intervention and protocol (e.g., ease of use, content, graphics). The findings will be used identify needs for any additional modifications to the intervention and protocol prior to the RCT.

ELIGIBILITY:
Aims 1 and 2 Only

Inclusion Criteria

Parents

1. Parents of patients of MMC Pediatrics aged 11-18
2. Refused HPV vaccination in the past two years
3. Have not received any doses of HPV vaccine
4. Own smartphone
5. Speak English
6. Have a clinic appointment scheduled within the coming month (AIM 1 Stage 2 & AIM 2 only)
7. Did not participate in Aim 1 Stage 1 (AIM 1 Stage 2 only)
8. Did not participate in Aim 1 Stage 1 or Aim 1 Stage 2 (Aim 2 only)

Providers

1. Physicians, physician assistants, and nurse practitioners who deliver primary care to patients aged 11-18 (Aim 1 Stage 1)
2. Physicians, physician assistants, and nurse practitioners who deliver primary care to patients aged 11-18 and the intervention at Meharry Medical College. (Aim 1 Stage 2, Aim 2)

Exclusion Criteria:

Parents

1. Parents with vaccinated patients or never been offered the vaccine in MMC pediatrics aged 11-18
2. Unvaccinated yet never refused the vaccine
3. Do not speak English
4. Do not own a smart phone
5. Does not have an upcoming clinic visit (Aim 1 Stage 2 and Aim 2)

Providers

1. Providers: Physicians, nurse practitioners, and physician assistants who do not deliver primary care to pediatric patients aged 11-18 at Meharry and other clinics
2. Providers who do not provide the HPV vaccine.
3. Providers who do not participate in Aim 1 stage 1 (Aim 1 Stage 2 only)
4. Did not pilot study (Aim 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | 6 months
  pre-screened, % contacted, % unable to contact, % screened, % enrolled, # enrolled per month
Retention Rates | 6 months
  % completed baseline survey, % came to clinic visit (primary retention endpoint), % completed post-visit survey
Data collection processes | 6 months
  % ascertained post-visit HPV vaccine status, # minutes to complete surveys

SECONDARY OUTCOMES:
HPV vaccine rates | 6 months
  # vaccinated post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No